CLINICAL TRIAL: NCT02590445
Title: Novel Deep Brain Stimulation in Ventral Capsule and Stratum for Refractory Obsessive-Compulsive Disorder: A Pilot Study
Brief Title: Novel Deep Brain Stimulation in Ventral Capsule and Stratum for Refractory Obsessive-Compulsive Disorder
Status: Unknown | Phase: Phase 2 / Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Ruijin Hospital (Other)
Responsible Party: Principal Investigator, Bomin Sun, Director of functional neurosurgery department, Ruijin Hospital
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Treatment
Other Study IDs: OCD pilot
Record Dates: First submitted 2015-10-26; First posted 2015-10-29 (Estimated); Last update posted 2016-12-06 (Estimated); Status verified 2016-12

CONDITIONS: Obsessive-Compulsive Disorder
MeSH Terms: conditions — Obsessive-Compulsive Disorder

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Active stimulation (Active Comparator): Stimulator on followed by off
  Interventions: Device: deep brain stimulation system
- Sham stimulation (Sham Comparator): Stimulator off followed by on
  Interventions: Device: deep brain stimulation system

INTERVENTIONS:
Device: deep brain stimulation system

SUMMARY:
Refractory obsessive-compulsive disorder (OCD) is a disabling condition. Deep brain stimulation (DBS) of ventral capsule/ventral striatum(VC/VS) is potentially the most effective treatment for refractory OCD. However, the affecting area of traditional electrodes is limited and not specific to VC/VS. The investigators designed a novel electrode, 2 mental contacts(3mm contact-2mm space-3 mm contact) could be implanted in ventral striatum and the other upper 2 contacts(4mm space-3mm contact-4mm space-3mm contact)that can be implanted in ventral capsule simultaneously, which the investigators believe will be more effective due to better compatibly with anatomical features of target area. This trial is to evaluate the effectiveness and safety of this approach.

ELIGIBILITY:
Inclusion Criteria:

1. Age between 18 and 65 years.
2. A primary diagnosis of OCD, defined according to the criteria of the Diagnostic and Statistical Manual of Mental Disorders, fifth edition (DSM-V).
3. Chronic: at least a 3-year history of OCD symptoms with psychosocial dysfunction
4. Severity: a score on the Yale-Brown Obsessive Compulsive Scale (Y-BOCS) of more than 25 or one subscale score of more than 15 ; a score for severity of illness on the Clinical Global Impression (CGI) scale of more than 4.
5. Disability: a score on the Global Assessment Functioning (GAF) scale of less than 45 or a score on Sheehan Disability Scale more than 24.
6. Refractory: a lack of response to drug therapy after adequate administration, defined as more than two types of serotonin reuptake inhibitors at the maximum tolerated dose for more than 12 weeks. Adequate behavior therapy, defined as more than 20 sessions psychotherapy with experienced therapist.
7. OCD medication regimen is stable for at least 4 weeks before enrollment.

Exclusion Criteria:

1. Schizophrenic disorder; bipolar disorder; substance abuse or dependence (except for dependence on nicotine), as assessed with the use of the Mini-International Neuropsychiatric Interview (MINI 6.0.0).
2. Cluster A or B personality disorder according to DSM-IV-TR criteria, as assessed with the use of the Structured Clinical Interview II.
3. A current severe major depressive episode, determined according to DSM-V criteria (as assessed with the use of the MINI 6.0.0) and defined by the Hamilton Depression Rating Scale-17 (HAMD) score of more than 20 and a risk of suicide.
4. Abnormal cognitive status (measured by MoCA), abnormal findings on functional magnetic resonance imaging (MRI) of the brain, or contraindications to surgery or anesthesia.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 8 (Estimated)
Dates: Start 2015-10; Primary Completion 2017-10 (Estimated); Study Completion 2018-04 (Estimated)

PRIMARY OUTCOMES:
Change in Yale-Brown Obsessive-Compulsive Scale (Y-BOCS) Score | Baseline (preoperative), 1 month, 3 months, 5 months, 6 months, 8 months, 12 months, 18 month, 24 month

SECONDARY OUTCOMES:
Change in Obsessive-Compulsive Inventory - Revised (OCI-R) Score | Baseline (preoperative), 1 month, 3 months, 5 months, 6 months, 8 months, 12 months, 18 month, 24 month
Adverse Events | Baseline (preoperative), 1 month, 3 months, 5 months, 6 months, 8 months, 12 months, 18 month, 24 month
Change in Hamilton Anxiety Scale, Hamilton Depression Scale-17 Score | Baseline (preoperative), 1 month, 3 months, 5 months, 6 months, 8 months, 12 months, 18 month, 24 month
Functional magnetic resonance imaging (fMRI) images | Baseline (preoperative)
Quality of life: Global assessment of function | Baseline (preoperative), 8 months, 12 months, 24 month
Disability: WHO disability assessment 2.0 | Baseline (preoperative), 8 months, 12 months, 24 month
Neurobehavior Task (Decision making task, such as Model task, IGT) | Baseline (preoperative), 8 months, 12 months, 24 month
Neurobehavior Task (Working memory task, such as N-back) | Baseline (preoperative), 8 months, 12 months, 24 month
Disability: Sheehan Disability Scale | Baseline (preoperative), 8 months, 12 months, 24 month
Change in Obsessional beliefs questionnaire (OBQ-44) Score | Baseline (preoperative), 1 month, 3 months, 5 months, 6 months, 8 months, 12 months, 18 month, 24 month
Change in Adult Temperament Questionnaire (ATQ-77) Score | Baseline (preoperative), 8 months, 12month, 24 month
Change in Temperament and Character Inventory Revised (TRI-R) Score | Baseline (preoperative), 8 months, 12month, 24 month
Cerebral glucose metabolism measured by PET-CT images | Baseline (preoperative), 12 month

CONTACTS AND LOCATIONS:
Overall Officials: Bomin Sun, MD, PhD, Principal Investigator — Ruijin Hospital
Locations (1):
- Shanghai Ruijin Hospital, Shanghai, Shanghai Municipality, China

REFERENCES:
- [Background] Goodman WK, Foote KD, Greenberg BD, Ricciuti N, Bauer R, Ward H, Shapira NA, Wu SS, Hill CL, Rasmussen SA, Okun MS. Deep brain stimulation for intractable obsessive compulsive disorder: pilot study using a blinded, staggered-onset design. Biol Psychiatry. 2010 Mar 15;67(6):535-42. doi: 10.1016/j.biopsych.2009.11.028. Epub 2010 Feb 8. PMID 20116047
- [Background] Mallet L, Polosan M, Jaafari N, Baup N, Welter ML, Fontaine D, du Montcel ST, Yelnik J, Chereau I, Arbus C, Raoul S, Aouizerate B, Damier P, Chabardes S, Czernecki V, Ardouin C, Krebs MO, Bardinet E, Chaynes P, Burbaud P, Cornu P, Derost P, Bougerol T, Bataille B, Mattei V, Dormont D, Devaux B, Verin M, Houeto JL, Pollak P, Benabid AL, Agid Y, Krack P, Millet B, Pelissolo A; STOC Study Group. Subthalamic nucleus stimulation in severe obsessive-compulsive disorder. N Engl J Med. 2008 Nov 13;359(20):2121-34. doi: 10.1056/NEJMoa0708514. PMID 19005196
- [Background] Denys D, Mantione M, Figee M, van den Munckhof P, Koerselman F, Westenberg H, Bosch A, Schuurman R. Deep brain stimulation of the nucleus accumbens for treatment-refractory obsessive-compulsive disorder. Arch Gen Psychiatry. 2010 Oct;67(10):1061-8. doi: 10.1001/archgenpsychiatry.2010.122. PMID 20921122